CLINICAL TRIAL: NCT02036359
Title: An Open-label, Randomized, Phase II Study of Erlotinib Monotherapy Versus Docetaxel and Cisplatin as Neoadjuvant Therapy in Patients of Stage IIIA Lung Adenocarcinoma With Epidermal Growth Factor Receptor Gene Mutation.
Brief Title: Erlotinib Monotherapy Versus Docetaxel and Cisplatin as Neoadjuvant Therapy in Patients of stageIIIA Lung ca
Acronym: Oncology
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201203009MIB
Record Dates: First submitted 2013-09-24; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
Keywords: Non-small Cell Lung Cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- erlotinib (Active Comparator): Patients in erlotinib arm will take erlotinib 150mg/day for 9 weeks unless disease progression, unacceptable toxicity or death.
  Interventions: Drug: erlotinib
- Chemotherapy (Active Comparator): Patients in chemotherapy arm will then receive 3 cycles (9 weeks) of chemotherapy with docetaxel 35mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 8.
  Treatment failure will include patients who fail to complete 3 cycles (9 weeks) of study treatments due to disease progression or unacceptable toxicity.
  Patients with no disease progression after terminating study treatment will undergo surgical resection and be followed until disease progression is noted, or study end. Survival will be recorded and analyzed.
  If progressive disease or unacceptable toxicity occurs during study treatments, patients will be treated at discretion of investigator according to local protocol.
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: erlotinib — 150mg/day for 9 weeks unless disease progression, unacceptable toxicity or death.
  Other Names: Tarceva
  Arms: erlotinib
Drug: docetaxel — receive 3 cycles (9 weeks) of chemotherapy with docetaxel 35mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 8.
  Other Names: Taxotere
  Arms: Chemotherapy

SUMMARY:
To compare clinical response (complete response and partial response) by RECIST) rates by RECIST between erlotinib monotherapy and docetaxel plus cisplatin chemotherapy

DETAILED DESCRIPTION:
an open-label, multi-centre, randomized, phase II study evaluating efficacy of erlotinib monotherapy vs. docetaxel plus cisplatin chemotherapy.

Patients with histological documented stage IIIA lung adenocarcinoma. The tumor specimens were examined for EGFR gene mutation (Exon 18-21).

Those with exon 19 deletion and L858R, G719X, L861Q mutation were randomized as erlotinib monotherapy or docetaxel plus cisplatin chemotherapy.

The randomization will be stratified by center

Study treatment Patients will receive treatment for 9 weeks unless disease progression, unacceptable toxicity or death.

Erlotinib arm:

Patients in erlotinib arm will take erlotinib 150mg/day for 9 weeks unless disease progression, unacceptable toxicity or death.

Chemotherapy arm:

Patients in chemotherapy arm will then receive 3 cycles (9 weeks) of chemotherapy with docetaxel 35mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 8.

Treatment failure will include patients who fail to complete 3 cycles (9 weeks) of study treatments due to disease progression or unacceptable toxicity.

Patients with no disease progression after terminating study treatment will undergo surgical resection and be followed until disease progression is noted, or study end. Survival will be recorded and analyzed.

If progressive disease or unacceptable toxicity occurs during study treatments, patients will be treated at discretion of investigator according to local protocol.

Please note:

• If it is judged by the investigator to be in the best interest of the patient, patients discontinuing study treatment may receive second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years, male or female

  * Able to comply with the protocol
  * Histologically documented stage IIIA lung adenocarcinoma
  * ECOG performance status 0-2
  * If the patient has the use coumarin (coumarin) (also to be called coumadin or warfarin), the patient applies drugs previous 7 days at the experiment to stop the medicine, and changes to other for to use the medicine.
  * Life expectancy > 12 weeks
  * Tumor specimen with EGFR gene mutation of exon 19 deletion and L858R, G719X, L861Q mutation
  * Adequate hematological function: ANC ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, Hb ≥ 9 g/dL
  * Data of INR and PTT should be available in patients taking anticoagulants concomitantly, with INR ≤ 1.5 and PTT ≤ 1.5 times the upper limit of normal (x ULN ) within 7 days prior to starting study treatment
  * Adequate liver function: serum bilirubin ≤ 1.5 x ULN; transaminases ≤ 2.5 x ULN
  * Adequate renal function: 24-hour urine creatinine clearance or creatinine clearance measured and calculated according to the formula of Cockroft and Gault ≥ 60ml/min
  * Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women
  * Written informed consent.
  * Patients are willing to complete FACT-L, ED-5Q, or pharmacoeconomic questionnaires

Exclusion Criteria:

* • Prior chemotherapy or treatment with another systemic anti-cancer agent (for example monoclonal antibody, tyrosine kinase inhibitor)

  * Mixed adenocarcinoma and other histological type of lung cancer
  * Unable to take oral medicine
  * Pregnant or lactating women
  * Fertile men or women of childbearing potential not using adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)
  * Malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, DCIS treated surgically with curative intent
  * Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to starting study treatment
  * Known hypersensitivity to any of the study drugs
  * Concurrent cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Event | Within 28 days of last study dose

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jen Yu, M.D., Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan